CLINICAL TRIAL: NCT06154018
Title: Heparin Reversal With Two Different Protamine Ratios After Cardiopulmonary By-pass.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Ioannina (Other)
Responsible Party: Principal Investigator, Evangelia Samara, Assistant Professor of Anesthesiology, University of Ioannina
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 179/23-2-2023
Record Dates: First submitted 2023-11-02; First posted 2023-12-01 (Actual); Last update posted 2024-05-31 (Actual); Status verified 2024-05

CONDITIONS: Cardiac Surgery; CAD; Valve Heart Disease; Coagulation Disorder
Keywords: cardiac surgery; heparin; protamin; coagulopathy; coagulopathy, viscoelastic tests
MeSH Terms: conditions — Heart Valve Diseases; Hemostatic Disorders | interventions — somatostatin, protamine zinc-

STUDY DESIGN:
Intervention Model Description: RCT
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 0.8:1 (Active Comparator): This arm will receive an initial administration of 0.8mg of protamine per 100IU of totally given heparin.
  Interventions: Drug: Protamin
- 0.6:1 (Active Comparator): This arm will receive an initial administration of 0.6mg of protamine per 100IU of totally given heparin.
  Interventions: Drug: Protamin

INTERVENTIONS:
Drug: Protamin — ACT and Clot- Pro test will be ran after initial and possible next protamine administrations
  Other Names: viscoelastic testing (Clot-Pro); ACT

SUMMARY:
Protamine is routinely used as a heparin reversal agent in cardiac surgery. However, its use may be associated with adverse events, while protamine excess may have additional anti-coagulant affect. Although guidelines advise towards a diminished reversal ratio, clinical practice remain heterogenic. The purpose of this study is to compare two different reversal ratios (0.6:1 και 0.8:1) of total heparin regarding the Activated Clotting Time (ACT), viscoelastic assays (Clot-Pro) and clinical hemorrhage.

A baseline ACT value and Clot Pro tests will be obtained prior to the operation start. After the initial reversal, ACT, Clot Pro tests will be conducted again. Coagulation factors are administrated according to Clot Pro results, and in case of ongoing clinical hemorrhage and any indication of heparin excess in the measured values, another 25mg of protamine is administrated, while tests are repeated.

DETAILED DESCRIPTION:
Protamine is routinely administered as a heparin-reversal factor in cardiac surgery. However, protamine is associated with specific adverse events, while it has additional anticoagulant effect while in excess. The literature supports that a reversal ratio lower than 1mg:100 IU (1:1) of heparin is safe and effective. According to recent studies, a ratio equal to 0.84:1 of initial or 0,6 of total heparin is safe and effective in cardiac surgery. Even lower ratios (<0,5:1) have been studied with positive outcomes.

The aim of this study is to evaluate the effectiveness of heparin reversal with two different protamin ratios (0,6:1 και 0,8:1) regarding the Activated Clotting Time (ACT), viscoelastic tests (Clot-Pro) and clinical hemorrhage.

Methods Perioperative management will follow standard department practice. The patients will be randomized to receive an initial dosage of protamine in a ratio 0.8 or 0.6 to 1 of the total heparin post cardiopulmonary by-pass disengagement. ACT and Clot Pro tests (IN, HI, EX and FIB-test) will run. In case of ongoing clinical hemorrhage, coagulation factors will administrated according to Clot Pro results, and in case of persistent clinical hemorrhage and any indication of heparin excess in the measured values, another 25mg of protamine will be administrated, while tests will be repeated. All patients will sign an informed consent prior to their inclusion in the study.

Data collection During pre-operative evaluation, age, weight, height, sex, BSA, ASA classification, Euroscore II, medication and co-morbidities will be documented.

Intraoperatively, anesthesia, cardiopulmonary bypass and aortic cross clamping time will be documented, as well as drugs administered and related adverse events.

Methods Induction in anesthesia will follow standard practice using fentanyl, prorofol and rocuronium. Maintenance will be achieved with sevoflurane. After induction in anesthesia and before heparin administration ACT and viscoelastic (Clot Pro) test results will be run using blood withdrawn form the patient's arterial line.

After disengagement from cardiopulmonary by-pass, protamine will be administered in a dosage according to randomization in a total volume of 60ml (diluted with normal saline). Five minutes later, another blood sample will be withdrawn form the patient's arterial line and ACT and Clot Pro tests (i.e. EX-, FIB-, IN- and HI- TEST) will be run again. In case of ongoing clinical bleeding, clotting factors will be administered according to the Clot PRo tests results. If bleeding persists, and there is and indication of either the ACT value or the IN to HI test ratio that there is heparin excess, another 25mg of protamine will be administered and ACT and Clot Pro tests will be repeated. The step can be repeated as many times as there is an indication of protamine excess and ongoing clinical bleeding. Transfusion and clotting products requirements will be recorded. Finally, the patients will be monitored for mechanical ventilation duration, transfusion requirements during ICU stay, postoperative bleeding and adverse events related to surgery and anesthesia for 48 hours postoperatively. A secondary analysis will depict the changes in thromboelastography before and after cardiopulmonary bypass as depicted in the ClotPro tests.

Purpose of the study The present study aims to evaluate two different ratios of heparin reversal (0.6 and 0.8 of total heparin)with protamine after the end of cardiopulmonary by pass in cardiac surgery patients. It is a prospective, randomized, comparative study of clinical hemorrhage, Activated Clotting Time (ACT) and viscoelastic tests using the ClotPro.Secondary endpoints are transfusion requirements, clotting factors administration, postoperative bleeding, mechanical ventilation duration and ICU length of stay.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Agreement to participate
* Scheduled for elective cardiac surgery on cardiopulmonary by-pass (CPB)

Exclusion Criteria:

* Age <18 years.
* No consent
* Known allergy to heparin or protamine
* History of Heparin Induced Thrombocytopenia (HIT)
* Off pump surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2023-03-18 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
Activated Clotting Time (in seconds) | Intraoperatively
  ACT values after heparin reversal
Viscoelastic testing | Intraoperatively
  CT-HI/CT-IN TEST values ratio after heparin reversal

SECONDARY OUTCOMES:
Transfusion | Intraoperatively and up to 24 hours postoperatively
  Number of blood products (RBC, FFP, PLT) administered to the patients
Clotting factors | Intraoperatively and up to 24 hours postoperatively
  Number of Clotting factors (PCCs, fibrinogen etc) administered to the patient
Postoperative hemorrhage | 24 hours postoperatively
  Total volume of blood drains and need for re-operation due to postoperative hemorrhage
ICU LOS | Up to 30 days
  Total ICU Length of Stay
Changes in ClotPro values in EX, FIB, IN and HI tests | intraoperatively
  differences in obtained values before and after cardiopulmonary bypass

CONTACTS AND LOCATIONS:
Overall Officials: Evangelia Samara, Md, PhD, Principal Investigator — University of Ioannina
Locations (1):
- University Hospital of Ioannina, Ioannina, Epirus, Greece

IPD SHARING:
Plan to Share IPD: No